CLINICAL TRIAL: NCT04595032
Title: MAnagement of METastatic Disease in Campania (MAMETIC): Role of Radiotherapy in an Italian Region: Protocol for an Observational Multicenter Trial
Brief Title: MAnagement of METastatic Disease in Campania (MAMETIC)
Acronym: MAMETIC
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: 33/20 oss
Record Dates: First submitted 2020-09-07; First posted 2020-10-20 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Disease
Keywords: Palliative care; Metastatic disease; Radiotherapy; Cancer pain; Breakthrough Cancer Pain; Quality of Life
MeSH Terms: conditions — Neoplasm Metastasis; Cancer Pain | interventions — Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: 3DCRT, IMRT, VMAT, SBRT — Radiation treatment

SUMMARY:
The MAMETIC Trial represents the first regional epidemiological study that aims to evaluate patients living in Campania with metastatic cancer, with the intent to detect different prevalence of tumors in the metastatic phase and evaluate the local response to the patient's request for assistance.

Condition or disease: Metastatic disease Intervention/treatment: Radiation Treatment

DETAILED DESCRIPTION:
The MAMETIC Trial is a multicenter, retrospective and prospective observational study and 17 of 20 RT Centers in Campania joined it.

1. The retrospective part of the study concerns all patients enrolled with a diagnosis of metastatic disease and treated in RT centers of the Campania Region with 3DCRT, IMRT, VMAT, SBRT techniques from January 2019 to August 2020. In 2019, it has been enrolled 12.500 patients in the 17 RT Centers and it is estimated that 20-30% of the above mentioned patients had metastasis. Thus, approximately 2.560 patients are expected to be enrolled.
2. The prospective part of the study is going to enroll all metastatic patients eligible for palliative RT, treated in RT Centers of the Campania region with 3DCRT, IMRT, VMAT, SBRT techniques from September 2020 to September 2025. Considering the RT Centers that joined the trial, it is expected to enroll approximately 2.500-4.200 patients per year and a total of 12.500-21.000 patients in 5 years.

The study will last 61 months, divided as follow: 60 months of enrollment phase and up to 1 month of follow-up for pain and bone metastasis patients. Follow-up will be performed on the 15th and 30th day after the end of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years resident in Campania Region;
* Patients diagnosed with metastatic disease candidates for radiotherapy
* Metastatic patients candidates for radiotherapy re-treatment
* Oligometastatic patients candidates for radiotherapy; Patients who have given their consent

Exclusion Criteria:

* Patients aged < 18 years
* Patients who are unable to express consent to sensitive data and radiant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic disease candidates for radiotherapy and resident in Campania region
Sampling Method: Non-Probability Sample
Enrollment: 3234 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Retrospective Study: Occurrence of palliative radiotherapy treatments in the Campania region | 20 months (Interval from January 2019 to August 2020)
  Occurrence of palliative radiotherapy treatments in the Campania region (Epidemiological Study)
Prospective Study: Occurrence of palliative radiotherapy treatments in the Campania region | 60 months (Interval from September 2020 to September 2025)
  Occurrence of palliative radiotherapy treatments in the Campania region (Epidemiological study)

SECONDARY OUTCOMES:
Retrospective Study: a. Incidence of metastatic disease at diagnosis | 20 months (Interval from January 2019 to August 2020)
  Incidence of metastatic disease at diagnosis
Retrospective Study: b. Time between first diagnosis and the onset of metastases | 20 months (Interval from January 2019 to August 2020)
  Time between first diagnosis and the onset of metastases
Prospective Study: Level A a. Incidence of metastatic disease at diagnosis | 60 months (Interval from September 2020 to September 2025)
  Incidence of metastatic disease at diagnosis
Prospective Study: Level A b. Time between first diagnosis and the onset of metastases | 60 months (Interval from September 2020 to September 2025)
  Time between first diagnosis and the onset of metastases
Prospective Study: Level A c. Interval from the first course of the radiation therapy to the retreatment | 60 months (Interval from September 2020 to September 2025)
  Interval from the first course of the radiation therapy to the retreatment (Epidemiological study)
Prospective Study: Level B a. Pain control | Up to 1 month after the end of RT
  Pain control measured for patient self-reporting of pain with Numeric Rating Scale (NRS) score, a 11-point scale (from 0 to 10), with higher scores indicating greater pain intensity
Prospective Study: Level C a. Quality of Life (QoL) according to European Organization for Research and Treatment of Cancer (EORTC) QLQ-C15-PAL questionnaire (health-related quality of life). | Until 2 weeks before RT
  Quality of life (QoL) according to European Organization for Research and Treatment of Cancer (EORTC) QLQ-C15-PAL questionnaire (health-related quality of life). It is scored on a metric from 0 to 10, higher scores mean better outcome
Prospective Study: Level C b. Functional performance measured by Palliative Performance Score (PPS). | Until 2 weeks before RT
  Functional performance measured by Palliative Performance Score (PPS). To score, there are 11 levels of PPS from 0% to 100% in 10 percent increments. Every decrease in 10% marks a fairly significant decrease in physical function.
Prospective Study: Level C c. Quality of life (QoL) of patients with bone metastases according to European Organization for Research and Treatment of Cancer (EORTC) QLQ-BM22 questionnaire (health-related quality of life). | Until 2 weeks before RT
  Quality of life (QoL) of patients with bone metastases according to European Organization for Research and Treatment of Cancer (EORTC) QLQ-BM22 questionnaire (health-related quality of life). It is scored on a metric from 0 to 100. Higher scores mean better outcome.
Prospective study: LEVEL C d. Incidence of spinal instability in patients with spinal metastases according to Spinal Instability Neoplastic Score (SINS) | Until 2 weeks before RT
  Incidence of spinal instability in patients with spinal metastases according to Spinal Instability Neoplastic Score (SINS). It is scored from 0 to 18. Higher scores mean worse outcome.
Prospective study: LEVEL C e. Evaluation of functional impairment as a result of their spinal cord injury according to the American Spinal Injury Association (ASIA) Score. | Until 2 weeks before RT
  Evaluation of functional impairment as a result of their spinal cord injury according to the American Spinal Injury Association (ASIA) Score. It is scored from 0 to 324. Higher scores mean better outcome.
Prospective study: LEVEL C f. Assessment of cognitive function in patients with brain metastases by Mini-Mental State Examination. | Until 2 weeks before RT
  Assessment of cognitive function in patients with brain metastases by Mini-Mental State Examination. It is scored from 0 to 30. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Muto, MD, Principal Investigator — National Cancer Institute of Naples
Locations (1):
- Radioterapia Oncologica INT IRCCS- Fondazione G.Pascale Sede Centrale, Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogenrieder T, Herlyn M. Axis of evil: molecular mechanisms of cancer metastasis. Oncogene. 2003 Sep 29;22(42):6524-36. doi: 10.1038/sj.onc.1206757. PMID 14528277
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Dillekas H, Demicheli R, Ardoino I, Jensen SAH, Biganzoli E, Straume O. The recurrence pattern following delayed breast reconstruction after mastectomy for breast cancer suggests a systemic effect of surgery on occult dormant micrometastases. Breast Cancer Res Treat. 2016 Jul;158(1):169-178. doi: 10.1007/s10549-016-3857-1. Epub 2016 Jun 15. PMID 27306422
- [Background] Gupta GP, Massague J. Cancer metastasis: building a framework. Cell. 2006 Nov 17;127(4):679-95. doi: 10.1016/j.cell.2006.11.001. PMID 17110329
- [Background] Dillekas H, Rogers MS, Straume O. Are 90% of deaths from cancer caused by metastases? Cancer Med. 2019 Sep;8(12):5574-5576. doi: 10.1002/cam4.2474. Epub 2019 Aug 8. PMID 31397113
- [Background] Huang JF, Shen J, Li X, Rengan R, Silvestris N, Wang M, Derosa L, Zheng X, Belli A, Zhang XL, Li YM, Wu A. Incidence of patients with bone metastases at diagnosis of solid tumors in adults: a large population-based study. Ann Transl Med. 2020 Apr;8(7):482. doi: 10.21037/atm.2020.03.55. PMID 32395526
- [Background] 7. AIOM-AIRTUM . Il numero del cancro in Italia 2019 . Intermedia Editore
- [Background] Coleman RE. Clinical features of metastatic bone disease and risk of skeletal morbidity. Clin Cancer Res. 2006 Oct 15;12(20 Pt 2):6243s-6249s. doi: 10.1158/1078-0432.CCR-06-0931. PMID 17062708
- [Background] Koswig S, Budach V. [Remineralization and pain relief in bone metastases after after different radiotherapy fractions (10 times 3 Gy vs. 1 time 8 Gy). A prospective study]. Strahlenther Onkol. 1999 Oct;175(10):500-8. doi: 10.1007/s000660050061. German. PMID 10554645
- [Background] Townsend PW, Smalley SR, Cozad SC, Rosenthal HG, Hassanein RE. Role of postoperative radiation therapy after stabilization of fractures caused by metastatic disease. Int J Radiat Oncol Biol Phys. 1995 Jan 1;31(1):43-9. doi: 10.1016/0360-3016(94)E0310-G. PMID 7995767
- [Background] Mirels H. Metastatic disease in long bones. A proposed scoring system for diagnosing impending pathologic fractures. Clin Orthop Relat Res. 1989 Dec;(249):256-64. PMID 2684463
- [Background] Chow E, Zeng L, Salvo N, Dennis K, Tsao M, Lutz S. Update on the systematic review of palliative radiotherapy trials for bone metastases. Clin Oncol (R Coll Radiol). 2012 Mar;24(2):112-24. doi: 10.1016/j.clon.2011.11.004. Epub 2011 Nov 29. PMID 22130630
- [Background] Sze WM, Shelley M, Held I, Mason M. Palliation of metastatic bone pain: single fraction versus multifraction radiotherapy - a systematic review of the randomised trials. Cochrane Database Syst Rev. 2004;2002(2):CD004721. doi: 10.1002/14651858.CD004721. PMID 15106258
- [Background] Di Franco R, Falivene S, Ravo V, Mammucari M, Sarli E, Baffini S, De Palma G, Pepe A, Traettino M, Muto M, Cappabianca S, Muto P. Management of painful bone metastases: our experience according to scientific evidence on palliative radiotherapy. Anticancer Res. 2014 Feb;34(2):1011-4. PMID 24511047
- [Background] Falivene S, Pezzulla D, Di Franco R, Giugliano FM, Esposito E, Scoglio C, Amato B, Borzillo V, D'Aiuto M, Muto P. Painful bone metastasis in elderly treated with radiation therapy: Single- or multiple-fraction regimen? A multicentre retrospective observational analysis. Aging Clin Exp Res. 2017 Feb;29(Suppl 1):143-147. doi: 10.1007/s40520-016-0671-x. Epub 2016 Nov 14. PMID 27844454
- [Background] 16. Giugliano FM, Di Franco R, Iadanza L, Borzillo V, Cutillo L and Muto P. Elderly Patients with Painful Bone Metastases. The Impact of Comorbidity on the Choice of Radiation Therapy Regimen. Journal of Palliative Care & Medicine
- [Background] 17. Di Franco R, Falivene S, Ravo V, Borzillo V, Giugliano FM, Argenone A, Rossetti S, Cavaliere C, D'aniello C, Romano FJ, Berretta M, Facchini G, Muto P. Impact of Procedural Pain In Radiotherapy Treatment WCRJ 2017; 4 (2): e884
- [Background] 18. Di Franco R, Calvanese M, Cuomo M, Manzo R, Murino P, Cappabianca S, Ravo V. Management of Painful Bone Metastases: The Interaction between Radiation Therapy and Zoledronate Journal of Cancer Therapy, 2011, 2, Published Online December 2011
- [Background] Kassam Z, Wong RK, Ringash J, Ung Y, Kamra J, DeBoer G, O'Brien M, Kim J, Loblaw DA, Wong S, Cummings B, Davey P. A phase I/II study to evaluate the toxicity and efficacy of accelerated fractionation radiotherapy for the palliation of dysphagia from carcinoma of the oesophagus. Clin Oncol (R Coll Radiol). 2008 Feb;20(1):53-60. doi: 10.1016/j.clon.2007.10.003. PMID 18345545
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Javed A, Pal S, Dash NR, Ahuja V, Mohanti BK, Vishnubhatla S, Sahni P, Chattopadhyay TK. Palliative stenting with or without radiotherapy for inoperable esophageal carcinoma: a randomized trial. J Gastrointest Cancer. 2012 Mar;43(1):63-9. doi: 10.1007/s12029-010-9206-4. PMID 20835926
- [Background] Rosenblatt E, Jones G, Sur RK, Donde B, Salvajoli JV, Ghosh-Laskar S, Frobe A, Suleiman A, Xiao Z, Nag S. Adding external beam to intra-luminal brachytherapy improves palliation in obstructive squamous cell oesophageal cancer: a prospective multi-centre randomized trial of the International Atomic Energy Agency. Radiother Oncol. 2010 Dec;97(3):488-94. doi: 10.1016/j.radonc.2010.09.001. Epub 2010 Oct 13. PMID 20950882
- [Background] Linskey ME, Andrews DW, Asher AL, Burri SH, Kondziolka D, Robinson PD, Ammirati M, Cobbs CS, Gaspar LE, Loeffler JS, McDermott M, Mehta MP, Mikkelsen T, Olson JJ, Paleologos NA, Patchell RA, Ryken TC, Kalkanis SN. The role of stereotactic radiosurgery in the management of patients with newly diagnosed brain metastases: a systematic review and evidence-based clinical practice guideline. J Neurooncol. 2010 Jan;96(1):45-68. doi: 10.1007/s11060-009-0073-4. Epub 2009 Dec 4. PMID 19960227
- [Background] Porceddu SV, Rosser B, Burmeister BH, Jones M, Hickey B, Baumann K, Gogna K, Pullar A, Poulsen M, Holt T. Hypofractionated radiotherapy for the palliation of advanced head and neck cancer in patients unsuitable for curative treatment--"Hypo Trial". Radiother Oncol. 2007 Dec;85(3):456-62. doi: 10.1016/j.radonc.2007.10.020. Epub 2007 Nov 26. PMID 18036689
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Sperduto PW, Berkey B, Gaspar LE, Mehta M, Curran W. A new prognostic index and comparison to three other indices for patients with brain metastases: an analysis of 1,960 patients in the RTOG database. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):510-4. doi: 10.1016/j.ijrobp.2007.06.074. Epub 2007 Oct 10. PMID 17931798
- [Background] Patil CG, Pricola K, Garg SK, Bryant A, Black KL. Whole brain radiation therapy (WBRT) alone versus WBRT and radiosurgery for the treatment of brain metastases. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD006121. doi: 10.1002/14651858.CD006121.pub2. PMID 20556764
- [Background] 28. Borzillo V, Giugliano FM, Di Franco R, Falivene S, Cammarota F, Ravo V, Muto P. Radiosurgery and Stereotactic Radiotherapy for Brain Metastases According the New Prognostic Indexes: our Preliminary Experience Neurol Neurophysiol 2015, 6:6
- [Background] Lam K, Zeng L, Zhang L, Tseng LM, Hou MF, Fairchild A, Vassiliou V, Jesus-Garcia R, Alm El-Din MA, Kumar A, Forges F, Chie WC, Sahgal A, Poon M, Chow E. Predictive factors of overall well-being using the EORTC QLQ-C15-PAL extracted from the EORTC QLQ-C30. J Palliat Med. 2013 Apr;16(4):402-8. doi: 10.1089/jpm.2012.0398. Epub 2013 Mar 4. PMID 23458649
- [Background] Yoon SJ, Choi SE, LeBlanc TW, Suh SY. Palliative Performance Scale Score at 1 Week After Palliative Care Unit Admission is More Useful for Survival Prediction in Patients With Advanced Cancer in South Korea. Am J Hosp Palliat Care. 2018 Sep;35(9):1168-1173. doi: 10.1177/1049909118770604. Epub 2018 Apr 16. PMID 29660991
- [Background] Mendez LC, Raman S, Wan BA, da Silva JLP, Moraes FY, Lima KMLB, Silva MF, Diz MDPE, Chow E, Marta GN. Quality of life in responders after palliative radiation therapy for painful bone metastases using EORTC QLQ-C30 and EORTC QLQ-BM22: results of a Brazilian cohort. Ann Palliat Med. 2017 Aug;6(Suppl 1):S65-S70. doi: 10.21037/apm.2017.04.06. Epub 2017 May 17. PMID 28595442
- [Background] van der Linden YM, Dijkstra SP, Vonk EJ, Marijnen CA, Leer JW; Dutch Bone Metastasis Study Group. Prediction of survival in patients with metastases in the spinal column: results based on a randomized trial of radiotherapy. Cancer. 2005 Jan 15;103(2):320-8. doi: 10.1002/cncr.20756. PMID 15593360
- [Background] Mizumoto M, Harada H, Asakura H, Hashimoto T, Furutani K, Hashii H, Takagi T, Katagiri H, Takahashi M, Nishimura T. Prognostic factors and a scoring system for survival after radiotherapy for metastases to the spinal column: a review of 544 patients at Shizuoka Cancer Center Hospital. Cancer. 2008 Nov 15;113(10):2816-22. doi: 10.1002/cncr.23888. PMID 18846565
- [Background] Shi DD, Hertan LM, Lam TC, Skamene S, Chi JH, Groff M, Cho CH, Ferrone ML, Harris M, Chen YH, Balboni TA. Assessing the utility of the spinal instability neoplastic score (SINS) to predict fracture after conventional radiation therapy (RT) for spinal metastases. Pract Radiat Oncol. 2018 Sep-Oct;8(5):e285-e294. doi: 10.1016/j.prro.2018.02.001. Epub 2018 Feb 13. PMID 29703703
- [Background] van Middendorp JJ, Goss B, Urquhart S, Atresh S, Williams RP, Schuetz M. Diagnosis and prognosis of traumatic spinal cord injury. Global Spine J. 2011 Dec;1(1):1-8. doi: 10.1055/s-0031-1296049. PMID 24353930
- [Background] Murray KJ, Scott C, Zachariah B, Michalski JM, Demas W, Vora NL, Whitton A, Movsas B. Importance of the mini-mental status examination in the treatment of patients with brain metastases: a report from the Radiation Therapy Oncology Group protocol 91-04. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):59-64. doi: 10.1016/s0360-3016(00)00600-3. PMID 10924972
- [Background] Dennis K, Linden K, Balboni T, Chow E. Rapid access palliative radiation therapy programs: an efficient model of care. Future Oncol. 2015;11(17):2417-26. doi: 10.2217/FON.15.153. Epub 2015 Aug 13. PMID 26271002
- [Background] Cellini F, Manfrida S, Deodato F, Cilla S, Maranzano E, Pergolizzi S, Arcidiacono F, Di Franco R, Pastore F, Muto M, Borzillo V, Donati CM, Siepe G, Parisi S, Salatino A, D'Agostino A, Montesi G, Santacaterina A, Fusco V, Santarelli M, Gambacorta MA, Corvo R, Morganti AG, Masiello V, Muto P, Valentini V. Pain REduction with bone metastases STereotactic radiotherapy (PREST): A phase III randomized multicentric trial. Trials. 2019 Oct 28;20(1):609. doi: 10.1186/s13063-019-3676-x. PMID 31661034
- [Derived] Di Franco R, Cascella M, Fusco M, Borzillo V, Scipilliti E, Ferraioli P, Iannacone E, De Palma G, Silvestro G, Gherardi F, Buonopane S, Alberti D, Totaro G, Manzo R, Guida G, Cuomo A, Pignata S, Di Napoli M, Rossetti S, Celentano E, Crispo A, Grimaldi M, Ravo V, Muto P. Management of Metastatic Disease in Campania (MAMETIC): An Observational Multicenter Retrospective and Prospective Trial on Palliative Radiotherapy in an Italian Region. Study Protocol. J Pain Res. 2022 Apr 8;15:1003-1010. doi: 10.2147/JPR.S336357. eCollection 2022. PMID 35422656